CLINICAL TRIAL: NCT04675476
Title: A Multilevel Intervention to Address Health Disparities in Lung Cancer Screening
Brief Title: A Patient and Provider Intervention to Address Health Disparities in Lung Cancer Screening
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY00003277
Record Dates: First submitted 2020-12-04; First posted 2020-12-19 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multilevel Intervention (Experimental)
  Interventions: Behavioral: Provider Prompt & Patient Outreach and Education
- Nonequivalent Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Provider Prompt & Patient Outreach and Education — To target lack of provider-prompted discussion about lung screening, an electronic medical record (EMR) message will be sent to primary care providers prior to scheduled visits with screening-eligible patients to notify them of the patient's eligibility and to encourage discussion of the benefits and limitations of the test. To target patient-level knowledge about lung screening, an outreach specialist will educate screening-eligible patients about the benefits and limitations of the test prior to their visit.
  Arms: Multilevel Intervention

SUMMARY:
To test the impact of a multilevel intervention on primary (provider-patient communication, intentions, and knowledge) and secondary (screening referrals and completion) outcomes.

DETAILED DESCRIPTION:
The proposed study will target two key levels of influence in the healthcare setting: provider and patient behavior in order to address disparities between African American and whites in lung screening awareness and utilization. Guided by NIH's Health Disparities Research Framework and building on the formative work conducted in the K99 phase, we will conduct a quasi-experimental study (pretest-posttest, with a nonequivalent control group) in partnership with four primary care clinics within the MedStar Health system in the R00 phase.

ELIGIBILITY:
Inclusion Criteria:

* 50-80 years old;
* current cigarette smoker or quit within 15 years;
* a 20+ pack-year smoking history;
* non-adherent to lung screening (>13 months);
* English-speaking;
* scheduled for an upcoming clinic appointment (4 weeks - 8 weeks); and
* able and willing to provide meaningful consent and complete telephone interviews

Exclusion Criteria:

* Individuals with a history of lung cancer

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
provider-patient discussion | 1-week post-visit
  Discussion about lung screening with the provider ('did you have a discussion with your doctor about lung screening?')
lung cancer screening intentions | 1-week post-visit
  Screening intentions ('how likely is it that you will undergo lung screening in the next 6-months?')
lung cancer screening knowledge | 1-week post-visit
  Lung cancer screening knowledge measure

SECONDARY OUTCOMES:
lung cancer screening referrals | 6-months
  Total number of lung screening orders captured via the electronic medical record
lung cancer screening completion rates | 6-months
  Total number of lung screening completions captured via the electronic medical record

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Health, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Williams RM, Whealan J, Sangraula A, Taylor KL, Adams-Campbell L, Miller KE, Glassmeyer K, Yee P, Camidge K, Foley K, Luta G, Lin KW, Barnes R, DuBoyce WF. Providing Reminders and Education Prior to lung cancer screening: Feasibility and acceptability of a multilevel approach to address disparities in lung cancer screening. Transl Behav Med. 2025 Jan 16;15(1):ibaf008. doi: 10.1093/tbm/ibaf008. PMID 40231692
- [Derived] Williams RM, Whealan J, Taylor KL, Adams-Campbell L, Miller KE, Foley K, Luta G, Brandt H, Glassmeyer K, Sangraula A, Yee P, Camidge K, Blumenthal J, Modi S, Kratz H. Multilevel approaches to address disparities in lung cancer screening: a study protocol. Implement Sci Commun. 2024 Feb 16;5(1):15. doi: 10.1186/s43058-024-00553-4. PMID 38365820